CLINICAL TRIAL: NCT01037816
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of FS-67 Patches in Adolescent Subjects With Ankle Sprain
Brief Title: FS-67 in the Treatment of Pediatric Patients With Ankle Sprain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hisamitsu Pharmaceutical Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FS-67-HP01-E02
Record Dates: First submitted 2009-12-18; First posted 2009-12-23 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Ankle Sprain
Keywords: Ankle Sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FS-67 patch (Active Comparator): One FS-67 patch applied to target ankle every 12 hours for three days (up to 6 FS-67 patches in three days)
  Interventions: Drug: FS-67 Patch
- Placebo Patch (Placebo Comparator): One placebo patch applied to target ankle every 12 hours for three days (up to 6 FS-67 patches in three days)
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: FS-67 Patch — One FS-67 patch applied to target ankle every 12 hours for three days (up to 6 FS-67 patches in three days)
  Other Names: Topical Patch
  Arms: FS-67 patch
Other: Placebo Patch — One placebo patch applied to target ankle every 12 hours for three days (up to 6 FS-67 patches in three days)
  Other Names: Sham treatment
  Arms: Placebo Patch

SUMMARY:
The objective of this study is assess the efficacy and safety of single and multiple applications of the FS-67 patch in the treatment of ankle sprain in pediatric population (ages 13-17).

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of FS-67 Patches in Adolescent Subjects With Ankle Sprain

ELIGIBILITY:
Inclusion Criteria:

* Grade 1 or Grade 2 ankle sprain

Exclusion Criteria:

* Pregnancy or lactation

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2009-12; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshinobu Higashi, Study Director — Hisamitsu Pharmaceutical Co., Inc.
Locations (22):
- United States (22):
  - Hisamitsu Investigator Site, Birmingham, Alabama
  - Hisamitsu Investigator Site, Tucson, Arizona
  - Hisamitsu Investigator Site, Hot Springs, Arkansas
  - Hisamitsu Investigator Site, Anaheim, California
  - Hisamitsu Investigator Site, Bell Gardens, California
  - Hisamitsu Investigator Site, Long Beach, California
  - Hisamitsu Investigator Site, Los Angeles, California
  - Hisamitsu Investigator Site, Boynton Beach, Florida
  - Hisamitsu Investigator Site, Daytona Beach, Florida
  - Hisamitsu Investigator Site, Doral, Florida
  - Hisamitsu Investigator Site, Jacksonville, Florida
  - Hisamitsu Investigator Site, Evansville, Indiana
  - Hisamitsu Investigator Site, Topeka, Kansas
  - Hisamitsu Investigator Site, Bellevue, Nebraska
  - Hisamitsu Investigator Site, Lincoln, Nebraska
  - Hisamitsu Investigator Site, Las Vegas, Nevada
  - Hisamitsu Investigator Site, Berlin, New Jersey
  - Hisamitsu Investigator Site, Charlotte, North Carolina
  - Hisamitsu Investigator Site, Columbus, Ohio
  - Hisamitsu Investigator Site, Dayton, Ohio
  - Hisamitsu Investigator Site, El Paso, Texas
  - Hisamitsu Investigator Site, Grapevine, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FS-67 Patch | Placebo Patch
Started | 126 | 126
Completed | 124 | 126
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FS-67 Patch | Placebo Patch | Total
Number analyzed (Participants) | 126 | 126 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 126 | 126 | 252
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 49 | 100
  Male | 75 | 77 | 152
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasians | 97 | 91 | 188
  Black or African American | 18 | 23 | 41
  Asians | 3 | 3 | 6
  European/Middle Eastern | 1 | 1 | 2
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Other | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 126 | 126 | 252

OUTCOME MEASURES:

1. Primary Outcome: Primary: Sum of Pain Intensity Difference (SPID) at 8-hours (SPID8) Upon Monopodal Weight Bearing.
Description: Summed Pain Intensity Differences (SPID8) worst observation carried forward (WOCF) during monopodal weight-bearing on the affected ankle observed at specified time-points (1, 2, 4, 6, & 8 hrs) after patch application. The SPID8 (WOCF) is a time-weighted sum of the pain intensity differences (PID), which were calculated as change from pain intensity at baseline to pain intensity at specified time points. Pain intensity was evaluated by means of a 100 mm visual analog scale (VAS), on which 0 mm represented no pain and 100 mm represented the worst pain imaginable. SPID8 was derived as the time-weighted sum (area under the curve) of the PID, where the weight assigned to each PID score is equal to the elapsed time (in hrs) since the previous scheduled evaluation time point. Five time-points were observed to calculate SPID8 therefore the potential SPID8 scores could range from -500 to +500 with negative values indicating increased pain over 8 hours.
Time Frame: 8 hours of patch application on Day 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FS-67 Patch | Placebo Patch
Number analyzed (Participants) | 126 | 126
units on a scale | 107.19 (9.05) | 89.13 (9.42)
Statistical Analysis 1: Comparison: FS-67 Patch vs Placebo Patch; The treatment effect of the FS-67 patch was estimated by computing the difference in LS means of the FS-67 and placebo patches from the ANCOVA model; Test type: Superiority; p = 0.137, ANCOVA

2. Secondary Outcome: Sum of Pain Intensity Difference at 8-hours (SPID8) at Rest.
Description: Summed Pain Intensity Differences (SPID8) worst observation carried forward (WOCF) at rest observed at specified time-points (1, 2, 4, 6, & 8 hrs) after patch application. The SPID8 (WOCF) is a time-weighted sum of the pain intensity differences (PID), which were calculated as change from pain intensity at baseline to pain intensity at specified time points. Pain intensity was evaluated by means of a 100 mm visual analog scale (VAS), on which 0 mm represented no pain and 100 mm represented the worst pain imaginable. SPID8 was derived as the time-weighted sum (area under the curve) of the PID, where the weight assigned to each PID score is equal to the elapsed time (in hrs) since the previous scheduled evaluation time point. Five time-points were observed to calculate SPID8 therefore the potential SPID8 scores could range from -500 to +500 with negative values indicating increased pain over 8 hours.
Time Frame: 8 hours of patch application on Day 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FS-67 Patch | Placebo Patch
Number analyzed (Participants) | 126 | 126
units on a scale | 111.98 (9.28) | 86.89 (9.65)
Statistical Analysis 1: Comparison: FS-67 Patch vs Placebo Patch; Test type: Superiority; p = 0.044, ANCOVA

ADVERSE EVENTS:
Time Frame: 3 day
Arm/Group | FS-67 Patch | Placebo Patch
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/126
Other Adverse Events (participants affected / at risk) | 14/126 | 15/126
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS-67 Patch (N=126) | Placebo Patch (N=126)
Application site reaction (General disorders) | 1 (2) | 4 (5)
Application site irritation (General disorders) | 2 (2) | 0 (0)
Application site erythema (General disorders) | 1 (1) | 1 (1)
Application site pruritus (General disorders) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No